CLINICAL TRIAL: NCT00535470
Title: An Open Label Study to Evaluate the Safety and Efficacy of Nitrogen Mustard (Mechlorethamine - MCH) 0.04% Formulation in Patients With Stage I-IIA Mycosis Fungoides Who Have Completed 12 Months Treatment Without a Complete Response
Brief Title: An Open Label Study to Evaluate the Safety and Efficacy of Mechlorethamine(MCH) 0.04% Formulation in Mycosis Fungoides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yaupon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007NMMF-202-US
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Open label 0.04% Mechlorethamine gel
  Interventions: Drug: 0.04% Mechlorethamine gel

INTERVENTIONS:
Drug: 0.04% Mechlorethamine gel — Mechlorethamine 0.04% PG applied to affected skin areas (lesions) once daily for up to seven (7) months. The frequency of application may be adjusted for toxicity. After seven (7) months, they will be terminated from the study.
  Other Names: Nitrogen Mustard 0.04%

SUMMARY:
To evaluate the efficacy and safety of topical application of MCH 0.04% in a propylene glycol ointment (PG)in patients with stage I or IIA MF previously treated with MCH 0.02% in a PG or AP ointment who did not achieve a complete response.

DETAILED DESCRIPTION:
This is a multi-center, open-label study of patients with previously treated stage I (IA and IB) or IIA MF who have not received a complete response after completing 12 months of treatment in clinical trial (2005NMMF-201-US)to either 0.02% MCH PG or 0.02% MCH in Aquaphor (AP) ointment formulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the treatment phase of the Yaupon Therapeutics-sponsored Phase II Pivotal study of MCH 0.02% in either the PG or AP formulation and have not achieved a complete response.

Exclusion Criteria:

* Pregnant or nursing females, or males and females of childbearing potential, not using an effective means of contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of topical application of NM 0.04% in a propylene glycol ointment (PG) in patients with stage I or IIA MF | 7 months

SECONDARY OUTCOMES:
Evaluate the tolerability and safety of topical application of NM 0.04% ointment formulations in patients with stage I or IIA MF | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lessin, M.D., Principal Investigator — Fox Chase Cancer Center
Locations (11):
- United States (11):
  - Stanford University Medical Center, Stanford, California
  - Northwestern University-Dept. of Dermatology, Chicago, Illinois
  - Columbia University, Dept of Dermatology, New York, New York
  - NYU Medical Center Dept. of Dermatology, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma University, Tulsa, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - The University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - Utah Clinical Trials, LLC, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Querfeld C, Scarisbrick JJ, Assaf C, Kim YH, Guitart J, Quaglino P, Hodak E. Chlormethine Gel Versus Chlormethine Ointment for Treatment of Patients with Mycosis Fungoides: A Post-Hoc Analysis of Clinical Trial Data. Am J Clin Dermatol. 2022 Jul;23(4):561-570. doi: 10.1007/s40257-022-00687-y. Epub 2022 May 10. PMID 35536441